CLINICAL TRIAL: NCT07069725
Title: A Phase 1, Open-label Positron Emission Tomography Trial to Assess Changes in Liver Uptake of [68Ga]Ga-FAPI-46 Following Oral Administration of Single Doses of AZD2389 to Patients With Advanced Liver Fibrosis (PECHORA).
Brief Title: The Phase 1, Open-label, PET Trial Designed to Investigate the Effect of AZD2389 on FAP Occupancy in the Liver in Participants With Advanced Liver Fibrosis.
Acronym: PECHORA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7930C00003
Record Dates: First submitted 2025-05-09; First posted 2025-07-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Liver Fibrosis; Hepatic Cirrhosis
Keywords: Liver Fibrosis; Hepatic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Positron-Emission Tomography

STUDY DESIGN:
Intervention Model Description: Groups of participants are assigned to receive interventions based on prior milestones being reached in the study, such as in some dose escalation and adaptive design studies.
Masking Description: This is an open-label trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part A (Other): In Part A, eligible participants (screening Visit 1) will return to the trial site for pre-assessments, confirmation of eligibility criteria, blood sampling for FAP concentration analysis (at the trial site), and the first PET examination (screening Visit 2). The participants will perform the PET examination at the PET Centre using the radioligand [68Ga]Ga-FAPI-46. Depending on the results of the initial PET examination, participants of Part A may be invited to continue the trial in Part B. In such a case they will participate in a total of 3 PET examinations, not exceeding predefined radiation exposure limits. If they do not participate further, they will complete the trial with a follow-up visit (Visit 3, telephone call) 7 days (±2 days) after the PET examination.
  Interventions: Diagnostic Test: PET scan and radioligand
- Part B1 (Experimental): In Part B1, eligible participants who completed the first PET scan at the screening visit and/or Part A will return to the trial site for blood sampling for FAP concentration analysis and the second PET examination on Day 1 (Visit 3) using the radioligand [68Ga]Ga-FAPI-46. At Visit 4, on Day 7 (±2 days), participants will receive a single oral dose of AZD2389. After AZD2389 administration, the third PET examination will be performed at the PET Centre followed by blood sampling for PK analysis and FAP activity, after which the participants will return to the trial site for further follow-up and safety monitoring. The participants will then be discharged from the trial site. Two follow up visits will occur after administration of AZD2389. Visit 5 (7 days [±2 days]) and Visit 6 (30 days[+7 days]) will monitor for safety and follow-up of AEs.
  Interventions: Drug: AZD2389; Diagnostic Test: PET scan and radioligand
- Part B2 (Experimental): In Part B2, eligible participants who completed the first PET scan at the screening visit and/or Part A will return to the trial site for blood sampling for FAP concentration analysis and the second PET examination on Day 1 (Visit 3) using the radioligand [68Ga]Ga-FAPI-46. At Visit 4, on Day 7 (±2 days), participants will receive a single oral dose of AZD2389. After AZD2389 administration, the third PET examination will be performed at the PET Centre followed by blood sampling for PK analysis and FAP activity, after which the participants will return to the trial site for further follow-up and safety monitoring. The participants will then be discharged from the trial site. Two follow up visits will occur after administration of AZD2389. Visit 5 (7 days [±2 days]) and Visit 6 (30 days[+7 days]) will monitor for safety and follow-up of AEs.
  Interventions: Drug: AZD2389; Diagnostic Test: PET scan and radioligand
- Part B3 (Experimental): In Part B3, eligible participants who completed the first PET scan at the screening visit and/or Part A will return to the trial site for blood sampling for FAP concentration analysis and the second PET examination on Day 1 (Visit 3) using the radioligand [68Ga]Ga-FAPI-46. At Visit 4, on Day 7 (±2 days), participants will receive a single oral dose of AZD2389. After AZD2389 administration, the third PET examination will be performed at the PET Centre followed by blood sampling for PK analysis and FAP activity, after which the participants will return to the trial site for further follow-up and safety monitoring. The participants will then be discharged from the trial site. Two follow up visits will occur after administration of AZD2389. Visit 5 (7 days [±2 days]) and Visit 6 (30 days[+7 days]) will monitor for safety and follow-up of AEs.
  Interventions: Drug: AZD2389; Diagnostic Test: PET scan and radioligand
- Part C (Experimental): In Part C (optional), participants attend the trial site during Visit 1 (screening, Day-35 to Day-14) to undergo an eligibility check. At Visit 2, the first PET examination with radioligand will be performed at least 5 days before IMP administration. At Visit 3 (Day 1), participants receive a single dose AZD2389, then undergo a second PET examination using the radioligand on Day 2, along with blood sampling for PK analysis and FAP activity. At Visit 4 (Day 8 ±2 days), participants will be admitted to the trial site for a second single dose, then undergo a third PET examination using the radioligand on Day 9, along with blood sampling. At Visit 5 (7 days ±2 days after the PET examination on Visit 4) and Visit 6 (30 days [+7 days]) after the drug administration on Visit 4), follow-up visits at the trial site take place for safety monitoring and follow-up of any AEs.
  Interventions: Drug: AZD2389; Diagnostic Test: PET scan and radioligand

INTERVENTIONS:
Drug: AZD2389 — Doses of AZD2389 will be administrated orally
  Arms: Part B1; Part B2; Part B3; Part C
Diagnostic Test: PET scan and radioligand — PET scan and radioligand
  Other Names: The participants will perform the PET examination at the PET Centre using the radioligand [68Ga]Ga-FAPI-46.

SUMMARY:
This is a phase 1, open-label, PET trial. The study is designed to investigate the effect of AZD2389 on FAP occupancy in the liver in participants with advanced liver fibrosis.

DETAILED DESCRIPTION:
This is a phase 1, open-label, PET trial in male and female patients with advanced liver fibrosis. The trial will consist of up to 3 sequential panels: Part A (Pilot panel), Part B (Main panel - 3 dose levels of AZD2389, 2 participants per dose level.), and Part C (optional panel). The design of the trial is adaptive and adjustments in time points and/or number of assessments and samples can be made during the course of the trial.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female (of non-childbearing potential) participant aged ≥ 20 years and willing and able to give written informed consent for participation in the trial.
2. History confirming compensated liver cirrhosis.
3. Females must have a negative pregnancy test.
4. Barrier contraceptives use by males.

Key Exclusion Criteria:

1. A condition that would interfere with evaluation of the trial intervention, put the participant at risk, influence the participant's ability to participate or affect the interpretation of the results of the trial.
2. Any clinically significant illness, medical or major surgical procedure or trauma prior randomization.
3. Hepatitis B , hepatitis C and/or HIV infection.
4. Significant elevations in liver blood test, MELD score >12 and platelets <100 x109/L g).
5. eGFR) < 60 ml/min/1.73m2.
6. History of decompensated liver cirrhosis.
7. Any participants with an aetiology of liver cirrhosis where the Investigator considers that PET signal uptake may be impacted.
8. History of bleeding disorders and major bleeding risk.
9. History of severe dermatological disorders or wound healing.
10. Positive screening result for drugs of abuse or alcohol.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Occupancy, %: percent change from baseline in uptake of FAP PET radioligand [68Ga]Ga-FAPI-46 in the liver after a single dose of AZD2389. | PART B: Day 7(+/-2 days); PART C: Day 2 and Day 8 (+/-2 days)
  To examine target FAP occupancy in the liver by AZD2389 as measured with [68Ga]Ga-FAPI-46 PET.

SECONDARY OUTCOMES:
Plasma concentrations of AZD2389. | PART B: Day 7(+/-2 days); PART C: Day 2 and Day 8 (+/-2 days)
  To evaluate plasma PK of AZD2389 after single doses.
AZD2389 PK parameters calculated by: the plasma concentration vs. time curve (AUC) from 0 to infinity (AUCinf) and maximum observed concentration (Cmax) | PART B: Day 7(+/-2 days); PART C: Day 2 and Day 8 (+/-2 days)
  Blood sampling and analysis to evaluate PK plasma of AZD2389 after single doses.
% FAP inhibition compared to baseline in plasma. | PART B: Day 7(+/-2 days); PART C: Day 2 and Day 8 (+/-2 days)
  To evaluate the plasma target engagement of AZD2389 by assessment of plasma FAP inhibition following single oral dosing.
% aTRV (for radioligand uptake). | PART B: Day 7(+/-2 days); PART C: Day 2 and Day 8 (+/-2 days)
  To quantify test-retest reproducibility of radioligand [68Ga]Ga-FAPI-46 uptake in the liver.
ICC (for radioligand uptake). | PART B: Day 7(+/-2 days); PART C: Day 2 and Day 8 (+/-2 days)
  To quantify test-retest reproducibility of radioligand [68Ga]Ga-FAPI-46 uptake in the liver.
Maximum possible target occupancy (Occmax). | PART B: Day 7(+/-2 days); PART C: Day 2 and Day 8 (+/-2 days)
  A theoretical relationship between average concentration of AZD2389 in plasma during the PET examination and radioligand binding will be assumed to calculate maximum target occupancy, if possible, by curve fitting.
The IC50 confidence interval | PART B: Day 7(+/-2 days); PART C: Day 2 and Day 8 (+/-2 days)
  A theoretical relationship between average concentration of AZD2389 in plasma during the PET examination and radioligand binding will be assumed to calculate the confidence interval associated with the IC50.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Research Site, Solna
  - Research Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/